CLINICAL TRIAL: NCT04273308
Title: The Effect of Whole-body Vibration Training on Biomarkers and Health Beliefs of Prefrail Older Adults: A Quasi-experimental Research
Brief Title: The Effect of Whole-body Vibration Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, HUI CHUN YANG, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201510ES014
Record Dates: First submitted 2019-11-06; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Biomarkers
Keywords: older adults; community; frailty biomarkers; health belief; prefrailty; quasi-experimental design; whole-body vibration training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- whole-body vibration training (Experimental): a 12-week whole-body vibration training that conducted 3 times per week, with 5-min continuous vibration at 12-Hz frequency and 3-mm amplitude each time.
  Interventions: Device: whole-body vibration training

INTERVENTIONS:
Device: whole-body vibration training — The experimental group participated in a 12-week whole-body vibration training that was conducted 3 times per week, with 5-min continuous vibration at 12-Hz frequency and 3-mm amplitude each time. The control group were provided home DVDs on resistance exercise and manuals for preventing frailty

SUMMARY:
The whole-body vibration programme employed in this study partly improved the biomarkers and health beliefs of the prefrail community-dwelling older adults.

DETAILED DESCRIPTION:
The experimental group participated in a 12-week whole-body vibration training that conducted 3 times per week, with 5-min continuous vibration at 12-Hz frequency and 3-mm amplitude each time

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years or older and living in a community
* Full consciousness and able to communicate verbally
* No severe cognitive disorder

Exclusion Criteria:

* Impaired mobility after recent surgery
* Major illness such as cancer
* Severe hearing impairment and inability to fully understand and follow instructions

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2016-06-25 (Actual); Study Completion 2016-06-25 (Actual)

PRIMARY OUTCOMES:
Pretest and posttest results of the experimental and control groups for Grip strength | Change from baseline at 12 weeks (The experimental group participated training that was conducted 3 times per week, with 5-min continuous vibration)
  Comparison of grip strength before and after 12 weeks of training
Pretest and posttest results of the experimental and control groups for 15-foot walk test speed | Change from baseline at 12 weeks (The experimental group participated training that was conducted 3 times per week, with 5-min continuous vibration)
  Comparison of 15-foot walk test speed before and after 12 weeks of training
Pretest and posttest results of the experimental and control groups for One-leg standing test using the dominant leg with the eyes open | Change from baseline at 12 weeks (The experimental group participated training that was conducted 3 times per week, with 5-min continuous vibration)
  Comparison of One-leg standing test with the eyes open before and after 12 weeks of training
Pretest and posttest results of the experimental and control groups for Thirty-second chair stand test | Change from baseline at 12 weeks (The experimental group participated training that was conducted 3 times per week, with 5-min continuous vibration)
  Comparison of Thirty-second chair stand test before and after 12 weeks of training
Pretest and posttest results of the experimental and control groups for Two-minute step test | Change from baseline at 12 weeks (The experimental group participated training that was conducted 3 times per week, with 5-min continuous vibration)
  Comparison of Two-minute step test before and after 12 weeks of training
Pretest and posttest results of the experimental and control groups for Health beliefs | The twelfth week
  Comparison of health beliefs before and after 12 weeks

SECONDARY OUTCOMES:
Summary of posttest ANCOVA of the experimental and control groups for biomarkers | The twelfth week
  One-way ANCOVA was conducted using the groups as the independent variable and the pretest results and sex as covariate variables to assess the intervention effectiveness
Summary of posttest ANCOVA of the experimental and control groups for health beliefs | The twelfth week
  One-way ANCOVA was conducted using the groups as the independent variable and the pretest results and sex as covariate variables to assess the intervention effectiveness